CLINICAL TRIAL: NCT01453894
Title: Center for Advancing Equity in Clinical Preventive Services Project 1: Improving Rates of Repeat Colorectal Cancer Screening
Brief Title: Improving Rates of Repeat Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Baker, Chief, Division of General Internal Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1P01HS021141-01-Project1; 1P01HS021141-01 (NIH)
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer Screening; Fecal Occult Blood Testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reminder and Outreach Intervention (Experimental): Participants randomized to this arm will receive the Reminder and Outreach intervention.
  Interventions: Behavioral: Reminder and Outreach Intervention
- Usual Care Control Group (No Intervention): Patients assigned to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Reminder and Outreach Intervention — This intervention includes (1) phone calls and text messages to remind participants that they are due for colorectal cancer (CRC) screening (2) mailed fecal occult blood test (FOBT) to participants so they can perform the test conveniently at home and mail them to the clinic, avoiding the need for a visit (3) plain language information and instructions to support understanding of CRC and FOBT use (4) a CRC screening coordinator to contact those still failing to complete testing by telephone or text (5) a feedback loop to patients regarding test results.
  Arms: Reminder and Outreach Intervention

SUMMARY:
The United States Preventive Services Task Force (USPSTF) recommends colorectal cancer (CRC) screening using fecal occult blood testing (FOBT), sigmoidoscopy, or colonoscopy in adults, beginning at age 50 and continuing until age 75. However, rates of CRC screening remain inadequate. In 2006, only 60.8% of adults 50 or older reported recent CRC screening. Screening rates are even lower among Black and Hispanic populations and in areas with higher poverty rates. Annual or biennial FOBT testing over many years is essential for FOBT to be effective. Few studies have examined the rate of repeat FOBT testing; to the investigators knowledge, none have been conducted in populations with high prevalence of barriers to screening (e.g., low literacy, varied cultural norms, and transportation difficulties). The assumption that FOBT is an effective CRC screening strategy presumes it will be done at least biennially, and cost-effectiveness studies of CRC screening strategies have found that the results are sensitive to the rate of adherence. The investigators study will provide critical information for providers and policymakers as they consider optimal strategies to increase CRC screening among vulnerable populations.

Overall Study Goal: Improve colorectal cancer screening by increasing rates of repeat fecal occult blood testing (FOBT).

Aim 1: Test if a multifaceted intervention increases repeat FOBT testing adherence over a 30-month period

Hypothesis 1: Compared to usual care, the intervention will increase the proportion of patients who complete a repeat annual FOBT within 6 months of their due date.

Hypothesis 2: Compared to usual care, the intervention will increase the proportion of patients who complete 2 additional FOBTs over the 30-month intervention period.

Aim 2: Explore perceived barriers to screening among patients who received the intervention but did not complete repeat FOBT testing within 18 months

Aim 3: Assess the costs of the intervention and the costs per additional repeat screening compared to patients who received usual care.

ELIGIBILITY:
Inclusion Criteria:

* Fecal occult blood test (FOBT) completed in the past year
* Age 51-75
* Preferred language English or Spanish

Exclusion Criteria:

* Any of the following: (1) Colonoscopy within 10 years (2) Flexible sigmoidoscopy within 5 years or (3) A clinician order or referral for FOBT prior to the due date
* Documentation of medical conditions suggesting colorectal cancer (CRC) screening through FOBT may be inappropriate including: chronic diarrhea, inflammatory bowel disease, iron deficiency, previous colonic polyp, use of medications in the previous 1 month that elevate the risk of a false-positive FOBT

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Baker, MD MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Baker DW, Brown T, Buchanan DR, Weil J, Balsley K, Ranalli L, Lee JY, Cameron KA, Ferreira MR, Stephens Q, Goldman SN, Rademaker A, Wolf MS. Comparative effectiveness of a multifaceted intervention to improve adherence to annual colorectal cancer screening in community health centers: a randomized clinical trial. JAMA Intern Med. 2014 Aug;174(8):1235-41. doi: 10.1001/jamainternmed.2014.2352. PMID 24934845
- [Derived] Baker DW, Brown T, Buchanan DR, Weil J, Cameron KA, Ranalli L, Ferreira MR, Stephens Q, Balsley K, Goldman SN, Wolf MS. Design of a randomized controlled trial to assess the comparative effectiveness of a multifaceted intervention to improve adherence to colorectal cancer screening among patients cared for in a community health center. BMC Health Serv Res. 2013 Apr 29;13:153. doi: 10.1186/1472-6963-13-153. PMID 23627550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients identified by query of electronic health record.
Period: Overall Study
Arm/Group | Reminder and Outreach Intervention | Usual Care Control Group
Started | 225 | 225
Completed | 225 | 225
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reminder and Outreach Intervention | Usual Care Control Group | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (6.1) | 59.6 (5.7) | 59.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 164 | 322
  Male | 67 | 61 | 128
Race/Ethnicity, Customized [Number; unit: participants]
  Latino/Hispanic | 197 | 205 | 402
  Other | 28 | 20 | 48
Region of Enrollment [Number; unit: participants]
  United States | 225 | 225 | 450
Insurance Status [Number; unit: participants]
  Uninsured | 174 | 172 | 346
  Insured | 51 | 53 | 104

OUTCOME MEASURES:

1. Primary Outcome: Completion of a Fecal Occult Blood Test (FOBT)
Description: This outcome will be categorized as Completed FOBT if a participant's chart has documentation of a completed FOBT screening test. Outcomes will be assessed by querying the electronic health record (EHR) for all participants.
Time Frame: within 6 months of randomization
Measure: Number; unit: participants
Arm/Group | Reminder and Outreach Intervention | Usual Care Control Group
Number analyzed (Participants) | 225 | 225
participants | 185 | 84

ADVERSE EVENTS:
Arm/Group | Reminder and Outreach Intervention | Usual Care Control Group
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/225
Other Adverse Events (participants affected / at risk) | 0/225 | 0/225

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No